CLINICAL TRIAL: NCT06152432
Title: Maxillary Implant Overdentures Retained by Bars or Locator Attachments: a 10-year Comparative Prospective Study.
Brief Title: Maxillary Implant Overdentures Retained by Bars or Locator
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18405
Record Dates: First submitted 2023-11-13; First posted 2023-11-30 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: Prospective comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxilillary implant overdenture retained by bars (Active Comparator): Patients treated with 4 dental implants in the edentulous maxilla and an overdenture retained by bars
  Interventions: Device: Maxillary implant overdenture
- Maxilillary implant overdenture retained by Locators (Active Comparator): Patients treated with 4 dental implants in the edentulous maxilla and an overdenture retained by solitary abutments (Locators)
  Interventions: Device: Maxillary implant overdenture

INTERVENTIONS:
Device: Maxillary implant overdenture — Patients with an edentulous maxilla and problems with their conventional denture are treated with an implant overdenture either retained by bars or Locators

SUMMARY:
* Background Patients experiencing problems with their conventional maxillary denture can benefit from implant- retained overdentures. Several retention systems are available. These retention systems can be roughly divided into bar-retained implant overdentures, in which multiple implants are splinted and the overdenture is attached through retentive clips, and into retention systems using non-splinted solitary attachments (locators). Evidence on maxillary implant overdenture attachment systems has been mostly short to medium term, non-comparing or retrospective. Even more, 10-years data of comparative studies are lacking.
* Main research question To compare treatment outcomes of fully edentulous patients with maxillary overdentures, supported by four implants, retained by either bars or locators . The primary objective of the study is to analyze marginal bone level changes by radiological assessments at 10-years follow-up. Secondary objectives are implant and overdenture survival, condition of peri- implant mucosa and patients' satisfaction.
* Design (including population, confounders/outcomes) The study design is an observational study of a group of patients which were treated 10 years ago with dental implants and an overdenture in the maxilla because of problems with retention and stability with their conventional denture. Outcomes: primary outcome is the change in marginal peri-implant bone level 10 years after placing the overdenture. Secondary outcome measures will be implant and overdenture survival, peri-implant mucosa health and patients' satisfaction using a questionnaire.

DETAILED DESCRIPTION:
• Introduction and rationale Patients experiencing problems with their conventional maxillary denture can benefit from implant-retained overdentures (IODs). Several retention systems are available. These retention systems can be roughly divided into bar-retained IODs, in which multiple implants are splinted and the overdenture is attached through retentive clips, and into retention systems using non-splinted solitary attachments. Bar-retained IOD's provide good retention, require little maintenance, but are more expensive than solitary attachments. Medium term results of bar-retained IODs are promising with high implant and overdenture survival and low incidence of complications and may be considered the gold standard. Solitary attachments serve as an alternative to bars. These attachments are more economical and are easy to clean by the patient, but wear more easily, which can cause lack of retention. However, replacement of these attachments can often be done chair side. A recent review reported that, when a maxillary IOD is supported by four implants, both types show equal implant survival, overdenture survival and patient satisfaction. However, these conclusions are based on a limited amount of randomized controlled trials. Moreover, most studies reporting on solitary attachments were retrospective. Evidence on maxillary IOD attachment systems has been mostly short to medium term, non-comparing or retrospective and therefore inconclusive. This underlines the need for studies comparing different attachment systems with a longer follow-up.

The study design is an observational study to compare treatment outcomes of fully edentulous patients with maxillary IODs, supported by four implants, retained by either bars or Locators. Patients were treated 10 years ago with dental implants and an overdenture in the maxilla because of problems with retention and stability with their conventional denture. Outcomes: primary outcome is the change in marginal peri-implant bone level 10 years after placing the overdenture. Secondary outcome measures will be implant and overdenture survival, peri-implant mucosa health and patients' satisfaction using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous patients or patients with an overdenture in the mandible, who were referred to the Department of Oral and Maxillofacial Surgery (University Medical Center Groningen, the Netherlands) 10 years ago, because they suffered from a lack of retention and stability of the upper (and lower) denture;
* Edentulous in the maxilla for at least one year;
* Sufficient bone volume in height in the anterior region of the maxilla to place the implants;
* The patient was 18 years or older;
* Sufficient interocclusal space for placement of an overdenture with attachment system;
* The patient was capable of understanding and giving informed consent.

Exclusion Criteria:

Exclusion criteria at the time of treatment:

* Patients with American Society of Anesthesiologists score (ASA score) ≥ III;
* Patients who were smoking;
* Patients with a history of radiotherapy in the head and neck region;
* Patients with a history of pre-prosthetic surgery or previous implant placement in the maxilla.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant marginal bone level | 10 years
  Difference in peri-implant bone level between start of functional period and at 10 years evaluation period

SECONDARY OUTCOMES:
Implant survival | 10 years
  Percentage of number of initially placed implants still in place after 10 years
Overdenture survival | 10 years
  Percentage of number of initially placed overdentures still in place after 10 years
Pocket probing depth | at 10 years
  Depth in millimeter of probing in the peri-implant sulcus
Plaque score | at 10 years
  Amount of plaque on implant abutment scored with the Modified Plaque Index, score 0-3, 3 is the worst
Peri-implant mucosa condition | at 10 years
  Health of peri-implant mucosa scored wit a Gingiva Index, score 0-3, 3 is the worst
Patient satisfaction | at 10 years
  Satisfaction of patients scored with a 5-point Likert scale, score 1-5, 5 is most dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Henny Meijer, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- Dept Oral and Maxillofacial Surgery UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No